CLINICAL TRIAL: NCT03357900
Title: Closed-loop Anaesthesia for Liver Transplantation: a Pilot Study
Acronym: THConcentr
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009/09; 2009-A00363-54 (Other: ANSM)
Record Dates: First submitted 2017-11-24; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Anesthesia; Liver Transplant
Keywords: Consciousness Monitor; Clinical Pharmacology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orthotopic liver transplantation (Experimental)
  Interventions: Device: Automated titration of propofol and remifentanil

INTERVENTIONS:
Device: Automated titration of propofol and remifentanil — Calculation of Consumption of propofol and remifentanil

SUMMARY:
Automated titration of propofol and remifentanil guided by the bispectral index (BIS) has been used for numerous surgical procedures. Orthotopic liver transplantation (OLT) uniquely combines major volaemic changes, an anhepatic phase, and ischaemia-reperfusion syndrome. We assessed the behaviour of this automated controller during OLT

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for OLT

Exclusion Criteria:

age younger than 18 years, pregnancy, allergy or hypersensitivity to propofol or remifentanil, a medical history of psychiatric illness, and supraspinal neurological disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-08-18 (Actual); Primary Completion 2012-02-09 (Actual); Study Completion 2012-02-09 (Actual)

PRIMARY OUTCOMES:
percentage of time spent in the BIS interval [40-60] | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No